CLINICAL TRIAL: NCT04904471
Title: A Global Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Clinical Trial to Evaluate the Efficacy, Safety, and Immunogenicity of Recombinant COVID-19 Vaccine (Sf9 Cells), for the Prevention of COVID-19 in Adults Aged 18 Years and Older
Brief Title: A Global Phase III Clinical Trial of Recombinant COVID- 19 Vaccine (Sf9 Cells)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: JSVCT109; NCT04887207 (obsolete NCT alias)
Record Dates: First submitted 2021-05-26; First posted 2021-05-27 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 Vaccine; Recombinant Vaccine; Efficacy; Safety; Immunnogenicity
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Three doses of recombinant SARS-CoV-2 vaccine (Sf9 Cell) on Day 0, Day 21and Day 42.
  Interventions: Biological: Recombinant COVID-19 vaccine (Sf9 cells)
- Placebo Comparator (Placebo Comparator): Three doses of placebo on Day 0, Day 21and Day 42.
  Interventions: Other: Placebo control

INTERVENTIONS:
Biological: Recombinant COVID-19 vaccine (Sf9 cells) — This vaccine is made by using baculovirus as a vector and expressing SARS-CoV-2 S-RBD in Sf9 cells, which is purified by antigen isolation and added with aluminum hydroxide adjuvant for the prevention of COVID-19.
  Arms: Experimental
Other: Placebo control — Except for the absence of study vaccine antigen, all other components (aluminum hydroxide, sodium chloride, sodium dihydrogen phosphate, disodium hydrogen phosphate) are consistent with the study vaccine and have been tested and qualified by National Institutes for Food and Drug Control.
  Arms: Placebo Comparator

SUMMARY:
This Phase III study is a global multicenter, randomized, double-blind,placebo controlled clinical trial to evaluate the efficacy, safety, and immunogenicity of therecombinant COVID-19 vaccine (Sf9 cells) in 40,000 participants aged 18 years and older who do not have a known history of SARS-CoV-2 infection but whose locations or circumstances put them at appreciable risk of acquiring COVID-19 or SARS-CoV-2 infection.

DETAILED DESCRIPTION:
This Phase III study is a global multicenter, randomized, double-blind, placebo-controlled clinical trial to evaluate the efficacy, safety, and immunogenicity of the recombinant COVID-19 vaccine (Sf9 cells) in 40,000 participants aged 18 years and older who do not have a known history of SARS-CoV-2 infection but whose locations or circumstances put them at appreciable risk of acquiring COVID-19 or SARS-CoV-2 infection. All participants will receive three doses of either study vaccine or placebo on Day 0, Day 21, Day 42 in a ratio of 1:1.There will be two cohorts in the study: the efficacy-safety cohort and the efficacy-extended safety-immunogenicity cohort. The efficacy will be evaluated in all vaccinated participants,including population in the efficacy-safety cohort, the efficacy-extended safety immunogenicity cohort. All vaccinated participants will also be followed up to monitor incidence of SAEs, MAAEs and AESIs. The reactogenicity of the vaccine will be evaluated in the efficacy-extended safety-immunogenicity cohort. Approximately 3000 participants will be enrolled into the efficacy-extended safety-immunogenicity cohort. This cohort will undergo additional visits to collect immunogenicity data associated with receiving the recombinant COVID-19 vaccine (Sf9 cells) and to analyze the infection status.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older.
* Able and willing (in the investigator's opinion) to comply with all study requirements.
* Willing to allow the investigators to discuss the volunteer's medical history with their general practitioner/personal doctor and access all medical records which are relevant to study procedures.
* Healthy adults, or stable-healthy adults who may have a pre-existing medical condition that does not meet any exclusion criteria. A stable medical condition is defined as a disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
* For females of childbearing potential only, willingness to practice continuous effective contraception (see glossary) for 90 days after completion of 3 doses vaccination, and have negative pregnancy tests before each dose vaccination. Note: Nonchildbearing potential is defined as surgically sterile (history of bilateral tubal ligation, bilateral oophorectomy, hysterectomy) or postmenopausal (defined as amenorrhea for ≥ 12 consecutive months prior to Screening without an alternative medical cause). A follicle-stimulating hormone (FSH) level may be measured at the discretion of the investigator to confirm postmenopausal status.
* Males participating in this study who are involved in heterosexual sexual activity must agree to practice adequate contraception (see glossary) and refrain from donating sperm for 90 days after receiving the study vaccination.
* Agreement to refrain from blood donation during the study.
* Provide a written informed consent form (ICF)

Exclusion Criteria:

Exclusion criteria for the first dose

* Participation in any other COVID-19 prophylactic drug trials during the duration of the study.

Note: Participation in COVID-19 treatment trials is allowed in the event of hospitalization due to COVID-19. The study team should be informed as soon as possible.

* Positive HIV antibody testing results.
* Participation in SARS-CoV-2 serological surveys where participants are informed of their serostatus during the duration of the study.

Note: Disclosure of serostatus post enrolment may accidentally unblind participants to group allocation. Participation in this trial can only be allowed if volunteers are kept blinded to their serology results from local/national serological surveys

* Planned receipt of any licensed or investigational vaccine, other than the study intervention,within 14 days before and after study vaccination.
* Prior receipt of an investigational or licensed COVID-19 vaccine.
* Administration of immunoglobulins and/or any blood products within three months prior to the planned administration of the investigational products (IPs).
* Any confirmed or suspected immunosuppressive or immunodeficient state; positive HIV status;asplenia; recurrent severe infections and chronic use (more than 14 days) of immunosuppressant medication within the past 6 months. Topical steroids or short-term (course lasting ≤14 days) oral steroids are not exclusion criteria.
* History of allergic disease or reactions likely to be exacerbated by any component of Recombinant COVID-19 Vaccine (Sf9 cells).
* Any history of angioedema
* Pregnancy, lactation, or willingness/intention to become pregnant within 90 days after receiving study vaccine
* Current diagnosis or treatment of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
* History of serious psychiatric condition likely to affect participation in the study
* A bleeding disorder (e g factor deficiency coagulopathy or platelet disorder) or prior history of significant bleeding or bruising following IM injections or venipuncture
* Suspected or known current alcohol or drug dependency
* Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease,liver disease, renal disease, an endocrine disorder, and neurological illness (mild/moderate well-controlled comorbidities are allowed)
* History of laboratory-confirmed COVID-19
* Continuous use of anticoagulants, such as coumarins and related anticoagulants (i.e. warfarin) or novel oral anticoagulants (i.e. apixaban, rivaroxaban, dabigatran, and edoxaban)
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study, or impair interpretation of the study data.

Exclusion criteria for the second/third dose In this trial, the second/third dose vaccination may be terminated in some cases. These include systemic allergic reactions, severe hypersensitivity reactions, or intolerable grade 3 or higher adverse reactions after the previous vaccination/placebo. If these reactions occur, the participants should not continue to receive the second/third vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39663 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Virologically confirmed (polymerase chain reaction(PCR) positive) symptomatic COVID-19 cases first occurring, regardless of severity. | 28 days after completion of 3 doses vaccination.
  Virologically confirmed (PCR positive) symptomatic COVID-19 cases first occurring ﹥ 28 days after completion of 3 doses vaccination, regardless of severity.
The incidence of serious adverse events(SAEs). | Day 0 to 6 months after completion of 3 doses vaccination.
  Serious adverse events(SAEs) from Day 0 through 6 months after completion of 3 doses vaccination.
The incidence of adverse event of special interests(AESIs). | Day 0 to 6 months after completion of 3 doses vaccination.
  Adverse event of special interests(AESIs) from Day 0 through 6 months after completion of 3 doses vaccination.
The incidence of medically attended adverse events(MAAEs). | Day 0 to 6 months after completion of 3 doses vaccination.
  Medically attended adverse events(MAAEs) from Day 0 through 6 months after completion of 3 doses vaccination.
The incidence of solicited adverse events(AEs). | 0 to 7 days after each dose vaccination
  Solicited adverse events(AEs) within 7 days after each dose vaccination.
The incidence of unsolicited adverse events(AEs) . | 0 to 21 days after the first dose and the second dose vaccination, and 0 to 28 days after the third dose vaccination
  Unsolicited adverse events(AEs) within 21 days after the first dose and the second dose, and within 28 days after the third dose vaccination.

SECONDARY OUTCOMES:
Virologically confirmed (polymerase chain reaction(PCR) positive) symptomatic COVID-19 cases first occurring , regardless of severity. | 14 days after completion of 3 doses vaccination.
  Virologically confirmed (polymerase chain reaction(PCR) positive) symptomatic COVID-19 cases first occurring ﹥14 days after completion of 3 doses vaccination, regardless of severity.
Severe COVID-19 and death (based on WHO criteria) caused by SARS-CoV-2 infection first occurring. | 14 days after completion of 3 doses vaccination.
  Severe COVID-19 and death (based on WHO criteria) caused by SARS-CoV-2 infection first occurring ﹥ 14 days after completion of 3 doses vaccination.
Severe COVID-19 and death (based on WHO criteria) caused by SARS-CoV-2 infection first occurring. | 28 days after completion of 3 doses vaccination
  Severe COVID-19 and death (based on WHO criteria) caused by SARS-CoV-2 infection first occurring ﹥ 28 days after completion of 3 doses vaccination.
Virologically confirmed (polymerase chain reaction(PCR) positive) hospitalised moderate, severe COVID-19 and death caused by SARS-CoV-2 infection first occurring. | 14 days after completion of 3 doses vaccination
  Virologically confirmed (polymerase chain reaction(PCR) positive) hospitalised moderate, severe COVID-19 and death caused by SARS-CoV-2 infection first occurring ﹥ 14 days after completion of 3 doses vaccination.
Virologically confirmed (polymerase chain reaction(PCR) positive) hospitalised moderate, severe COVID-19 and death caused by SARS-CoV-2 infection first occurring. | 28 days after completion of 3 doses vaccination
  Virologically confirmed (polymerase chain reaction(PCR) positive) hospitalised moderate, severe COVID-19 and death caused by SARS-CoV-2 infection first occurring ﹥ 28 days after completion of 3 doses vaccination.
Serologically confirmed SARS-CoV-2 infection or virologically confirmed (polymerase chain reaction(PCR) positive) COVID-19 cases first occurring, regardless of symptomatology or severity. | 14 days after completion of 3 doses vaccination
  Serologically confirmed SARS-CoV-2 infection or virologically confirmed (polymerase chain reaction(PCR) positive) COVID-19 cases first occurring ﹥ 14 days after completion of 3 doses vaccination, regardless of symptomatology or severity.
Serologically confirmed SARS-CoV-2 infection or virologically confirmed (polymerase chain reaction(PCR) positive) COVID-19 cases first occurring, regardless of symptomatology or severity. | 28 days after completion of 3 doses vaccination
  Serologically confirmed SARS-CoV-2 infection or virologically confirmed (polymerase chain reaction(PCR) positive) COVID-19 cases first occurring ﹥ 28 days after completion of 3 doses vaccination, regardless of symptomatology or severity.
The incidence of serious adverse events(SAEs) in all participants. | Day 0 to 12 months after completion of 3 doses vaccination
  Serious adverse events(SAEs) from Day 0 through 12 months after completion of 3 doses vaccination in all participants.
The incidence of medically attended adverse events(MAAEs) in all participants. | Day 0 through 12 months after completion of 3 doses vaccination
  Medically attended adverse events(MAAEs) from Day 0 through 12 months after completion of 3 doses vaccination in all participants.
The incidence of adverse event of special interests(AESIs) in all participants. | Day 0 through 12 months after completion of 3 doses vaccination
  Adverse event of special interests(AESIs) from Day 0 through 12 months after completion of 3 doses vaccination in all participants.
The geometric mean increase(GMI) of specific antibody. | Day 28, month 3, month 6, and month 12 after completion of 3 doses vaccination
  The geometric mean increase(GMI) of spike protein (S) receptor binding domain RBD region(S-RBD) IgG antibody on day 28, month 3, month 6 and month 12 after completion of 3 doses vaccination, measured by enzyme-linked immunosorbent assays(ELISA).
The seroconversion rate of specific antibody. | Day 28, month 3, month 6, and month 12 after completion of 3 doses vaccination
  The seroconversion rate of spike protein (S) receptor binding domain RBD region(S-RBD) IgG antibody on day 28, month 3, month 6 and month 12 after completion of 3 doses vaccination, measured by enzyme-linked immunosorbent assays(ELISA).
The geometric mean titer(GMT) of specific antibody. | Day 28, month 3, month 6, and month 12 after completion of 3 doses vaccination
  The geometric mean titer(GMT) of spike protein (S) receptor binding domain RBD region(S-RBD) IgG antibody on day 28, month 3, month 6 and month 12 after completion of 3 doses vaccination, measured by enzyme-linked immunosorbent assays(ELISA).
The seroconversion rate of live-virus neutralizing antibody. | Day 28, month 3, month 6, and month 12 after completion of 3 doses vaccination
  The seroconversion rate of live-virus neutralizing antibody on day 28, month 3, month 6 and month 12 after completion of 3 doses vaccination.
The geometric mean titer(GMT) of live-virus neutralizing antibody. | Day 28, month 3, month 6, and month 12 after completion of 3 doses vaccination
  The geometric mean titer(GMT) of live-virus neutralizing antibody on day 28, month 3, month 6 and month 12 after completion of 3 doses vaccination.
The geometric mean increase(GMI) of live-virus neutralizing antibody. | Day 28, month 3, month 6, and month 12 after completion of 3 doses vaccination
  The geometric mean increase(GMI) of live-virus neutralizing antibody on day 28, month 3, month 6 and month 12 after completion of 3 doses vaccination.

OTHER OUTCOMES:
SARS-CoV-2 virus nucleic acid sequence of COVID-19 cases that occurred derived from isolates or direct NP/OP swab. | 28 days after completion of 3 doses vaccination
  SARS-CoV-2 virus nucleic acid sequence of COVID-19 cases that occurred > 28 days after completion of 3 doses vaccination derived from isolates or direct NP/OP swab.
Virologically confirmed (polymerase chain reaction(PCR) positive) symptomatic COVID-19 cases first occurring in different age groups, regardless of severity. | 28 days after completion of 3 doses vaccination
  Virologically confirmed (polymerase chain reaction(PCR) positive) symptomatic COVID-19 cases first occurring ﹥28 days after completion of 3 doses vaccination in different age groups (18-59 group and ≥60 groups), regardless of severity.

CONTACTS AND LOCATIONS:
Locations (24):
- Indonesia (6):
  - Puskesmas Ciketingudik, Bekasi, Jiangsu
  - Permata Hospital, Bekasi
  - Brawijaya University Hospital, Malang
  - Universitas Muhammadiyah Malang Hospital, Malang
  - Airlangga University Hospital, Surabaya
  - Husada Utama Hospital, Surabaya
- Kenya (2):
  - Moi Teaching and Referral Hospital，Eldoret (MTRH), Eldoret
  - KAVI-Institute of Clinical Research, University of Nairobi, Nairobi
- Mexico (7):
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Centro de Investigación Clínica y medicina traslacional (CIMeT), Guadalajara
  - Hospital General Dr. Manuel Gea González, Mexico City
  - Invesclinic MX, Mexico City
  - Clínica de Enfermedades Crónicas y de Procedimientos Especiales, Morelia
  - SMIQ，S de R.L. de C.V., Querétaro
  - FS Scientia Pharma SA de CV, San Luis Potosí City
- Bharatpur Hospital, Kathmandu, Nepal
- Philippines (8):
  - Perpetual Succour Hospital - The Research Institute, Cebu City
  - St Luke Medical Centre - BGC, City of Taguig
  - De La Salle Medical and Health Sciences Institute, Dasmariñas
  - The Medical City - Iloilo, Iloilo City
  - West Visayas State University Medical Center, Iloilo City
  - Tropical Disease Foundation, Makati City
  - Makati Medical Center, Makati City
  - Quirino Memorial Medical Center, Quezon City